CLINICAL TRIAL: NCT05786339
Title: Bioequivalence Study of Two Irbesartan in Healthy Chinese Subjects: an Open, Randomized, Single-Dose and Crossover Study
Brief Title: Bioequivalence Study of Two Irbesartan in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SZHB17-007
Record Dates: First submitted 2023-02-03; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Therapeutic Equivalency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference formulation (Experimental): Irbesartan tablet (0.15g/tablet) , Manufacturer: Sanofi Clir SNC
  Interventions: Drug: Reference Irbesartan Tablet
- Test formulation (Experimental): Irbesartan tablet (0.15g/tablet) , Manufacturer: Shenzhen Haibin Pharmaceutical Co., Ltd.
  Interventions: Drug: Tested Irbesartan Tablet

INTERVENTIONS:
Drug: Tested Irbesartan Tablet — T
  Arms: Test formulation
Drug: Reference Irbesartan Tablet — R
  Arms: Reference formulation

SUMMARY:
The bioavailability of Irbesartan (150 mg) developed by Shenzhen Haibin Pharmaceutical Co., Ltd. was compared with that of reference Irbesartan (Aprovel ®,150 mg) produced by Sanofi Clir SNC. The bioequivalence of single dose of test preparation and reference preparation was evaluated in heathy subjects under fasting and fed conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female aged over 18years
2. Subjects willing to provide written informed consent and to adhere to protocol requirements
3. Subject's weight within normal range according to normal values for Body Mass Index (19.00 to 26.00 kg/m2 (both inclusive)), males with minimum of 50 kg weight, females with minimum of 45kg weight.
4. Subjects have not clinically significant abnormalities, including vital signs, physical examinations, laboratory tests, and ECG as determined by clinical examination

Exclusion Criteria:

1. History or presence of significant cardiovascular, Urogenital, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder
2. Allergic constitution(Allergic to two or more substances) or hypersensitivity to investigational product
3. History or presence of significant gastrointestinal inflammation /ulcer. or other medical history affecting drug absorption
4. Use of any drugs or herbal medicine within 14 days prior to the first dose
5. Can not follow approved birth control methods (a double barrier method) from the screening（Female subjects from two weeks prior to the screening） till 3 months after the last dose -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-11-17 (Actual); Primary Completion 2019-01-16 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Cmax | 48hours
  Evaluation of Peak Plasma Concentration
AUC0-t | 484hours
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-t
AUC0-∞ | 48hours
  Evaluation of Area under the plasma concentration versus time curve

SECONDARY OUTCOMES:
safety | 30days
  Monitor all the adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Yu Cao, Principal Investigator — The Affiliated Hosptial of Qingdao University
Locations (1):
- Affiliated Hospital of Qingdao University Phase I Clinical Research Center, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No